CLINICAL TRIAL: NCT02893969
Title: Multicentre, Randomized Clinical Trial of Pediatric Concussion Assessment of Rest and Exertion (PedCARE): A Study to Determine When to Resume Physical Activities Following Concussion in Children
Brief Title: Pediatric Concussion Assessment of Rest and Exertion
Acronym: PedCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Ontario Spor Support Unit (Other); Holland Bloorview Kids Rehabilitation Hospital (Other); Western University, Canada (Other); The Hospital for Sick Children (Other); Children's Hospital of Western Ontario (Other)
Responsible Party: Principal Investigator, Roger Zemek, Associate Professor, Dept. of Pediatrics and Emergency Medicine, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/80X
Record Dates: First submitted 2016-08-02; First posted 2016-09-09 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Concussions; Post-Concussive Symptoms
Keywords: Physical Activity; Rest
MeSH Terms: conditions — Post-Concussion Syndrome; Motor Activity | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Gradual reintroduction of non-contact physical activity at 72 hours post-concussion.
  Interventions: Behavioral: Physical Activity
- Control Group (Sham Comparator): Physical and cognitive rest post-injury until fully asymptomatic. Once asymptomatic participants can gradually reintroduce physical activity.
  Interventions: Behavioral: Rest

INTERVENTIONS:
Behavioral: Physical Activity — After 72 hours of full physical rest patients will gradually reintroduce physical activity into their daily routine.
  Arms: Experimental group
Behavioral: Rest — Complete physical rest until asymptomatic.
  Arms: Control Group

SUMMARY:
The goal of this study is to investigate when is the best time to resume physical activity following a head injury. Two treatment plans will be studied; the first treatment plan consists of gradually reintroducing physical activity in the child's routine, starting 72 hours following the head injury. The second treatment plan involves physical and mental rest until the child as no more symptoms. Once symptom free, physical activity is gradually reintroduced in the child's routine.

DETAILED DESCRIPTION:
Persistent post-concussive symptoms (PPCS) pose long-term challenges and can impact negatively patients' health-related quality of life and functional outcomes. Preventing PPCS, pediatric concussion guidelines call for cognitive and physical rest. Strict physical activity restriction is recommended until symptom-free, followed by a progressive step-wise return to activities. Unfortunately, little evidence beyond expert opinion exists to guide health care professionals on how and when to best re-introduce physical activity to hasten recovery and reduce the burden of PPCS. Recent evidence suggests protracted rest may hinder recovery. In fact, early resumption of physical exercise has proven physiological, psychological and functional benefits in many other conditions, including stroke (a severe traumatic brain injury). Findings from pilot studies in children with PPCS support that early, active rehabilitation is associated with improved recovery.

The goal of this study is to investigate whether early reintroduction of non-contact, physical activity at 72-hour post-injury reduces the rate of PPCS in children following an acute concussion as compared to usual care stepwise resumption of activity only once fully asymptomatic as per the Zurich consensus return-to-play protocol.

The study is a multicentre, blind, randomized clinical trial. A total of 350 participants will be recruited from 3 Pediatric Emergency Research Canada (PERC) Emergency Departments (ED). Eligible children are those aged 10-17 years who sustained a concussion in the previous 48 hours. Participants will be randomized to either the experimental intervention group or the the control group. The experimental intervention group consist of resumption of light, aerobic exercise (e.g., 15 minute walk) 72 hours post-injury, irrespective of symptoms. Patients will be allowed to progress activity daily using one of the following of their choice: Frequency, Intensity, Time (duration), or Type, as long as symptoms are well-tolerated, with a minimum of 24 hours between each step. Control group: Usual care according to Zurich return-to-play guidelines (complete rest until full resolution of concussion symptoms [several weeks of rest may be required prior to initiation], followed by stepwise activity progression).

ELIGIBILITY:
Inclusion Criteria:

Subjects presenting to one of the study hospital EDs after sustaining a direct or indirect head injury will be eligible if they:

* aged 10 through 17.99 years;
* have a concussion, defined by Zurich consensus statement;
* suffered the initial injury in the previous 48 hours;
* are proficient in English or French.

Exclusion Criteria:

Patients will be excluded if they present with traumatic head injuries with any of the following:

* Glasgow Coma Scale ≤13;
* abnormality on standard neuroimaging studies, including positive head CT findings (Note: neuroimaging is not required, but may be performed if clinically indicated);
* neurosurgical operative intervention, intubation or intensive care required;
* multi-system injuries with treatment requiring hospital admission, operating room or procedural sedation in ED (Note: hospital admission for observation or management of ongoing concussion symptoms is not an exclusion criteria);
* severe chronic neurological developmental delay resulting in communication difficulties; intoxication at the time of ED presentation as per clinician judgment;
* no clear history of trauma as primary events (e.g., seizure, syncope or migraine);
* inability to resume physical activities (e.g., fractured extremity or other concomitant injuries);
* inability to obtain a proper written informed consent/assent (language barrier, absence of parental authority, developmental delay, intoxication, patient too confused to consent, etc.);
* legal guardian not present (certain forms need be completed by parents/legal guardians).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 456 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Health and Behaviour Inventory (HBI) | 2 weeks
  The HBI is a 20-item self-report questionnaire, Likert scale (0, 1, 2, or 3 points) yielding separate scores for cognitive and somatic symptom scales for a total score range of 0 to 60

SECONDARY OUTCOMES:
Post-Concussion Symptom Inventory (PCSI) | 2 and 4 weeks
  Post-Concussion Symptom Inventory (PCSI) will be used as a confirmatory instrument for defining a PPCS case. PCSI is a validated, comprehensive self-administered instrument that has been used in other pediatric concussion studies, and only one of two measures applicable to younger children with published validity and reliability data. For the purpose of this study the investigators will be using the PCSI pre-adolescent scale version (18-item, 3-point scale), encompassing physical, cognitive, emotional and sleep domains. The scale will be used for all the children in the study. This specific version has demonstrated excellent internal consistency (r=0.87 for children aged 8-12 years). The assessment will be included in the second and fourth week follow-ups.
The Pediatric Quality of Life Inventory™ version 4.0 (PedsQL-4.0) | 2 and 4 weeks
  The PedsQL is a reliable and valid measure of health-related quality of life in healthy children and adolescents and those with acute and/or chronic health conditions.120 Parent versions exist for children aged 2 to 18 years (in 4-age groups) and child versions for those aged 5 and over. For this study only the child's version (ages 8-12 (appendix 16a) and ages 13-18 (appendix 16b)) will be used. The inventory covers four domains: physical, emotional, social and school and takes approximately 4 minutes to complete. The 18-item PedsQL™ Multidimensional Fatigue Scale is designed to measure fatigue in pediatric patients and comprises the General Fatigue Scale (6 items), Sleep-Rest Fatigue Scale (6 items), and Cognitive Fatigue Scale (6 items). The PedsQL™ Multidimensional Fatigue Scale has demonstrated excellent internal consistency reliability and validity. For the purpose of this study only the child version will be administered during the 2 and 4th week follow-up.
Pediatric Injury Functional Outcome Scale (PIFOS) | 2 and 4 weeks
  The PIFOS is an assessment that evaluates functional outcomes. The PIFOS is a 26-item structure interview, and is completed by caregivers. The assessment elicits ratings regarding motor skills, daily living skills, communication skills, cognition, social-emotional functioning, physical changes, and academic functioning.
14 days physical activity monitoring with an Actical watch z-model | 2 weeks
  The Actical will provide an objective measurement of activity/sedentary monitoring. The device is capable of encoding raw acceleration, activity counts, energy expenditure, physical activity intensity, body position, and amount of sleep. The device can store up to 32 MB data (194 days on the Epoch mode of 1 second) and the battery provides power for 180 days between charges. The Acticsl has been validated and is a reliable measure.
Patients long-term health-care utilization (e.g. what health care services patient access) and risks for concussion-related comorbidities, data will be collected through the Institute for Clinical Evaluative Sciences (ICES) data linkage. | 20 years
  Investigating the long-term health-care utilization of concussion patients and determining the risks for concussion-related comorbidities will be done with ICES data linkage.

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Zemek, MD, Principal Investigator — CHEO
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledoux AA, Barrowman NJ, Boutis K, Davis A, Reid S, Sangha G, Farion KJ, Belanger K, Tremblay MS, Yeates KO, DeMatteo C, Reed N, Zemek R; Pediatric Emergency Research Canada PedCARE team. Multicentre, randomised clinical trial of paediatric concussion assessment of rest and exertion (PedCARE): a study to determine when to resume physical activities following concussion in children. Br J Sports Med. 2019 Feb;53(3):195. doi: 10.1136/bjsports-2017-097981. Epub 2017 Jul 12. PMID 28701360
- [Derived] Ledoux AA, Barrowman N, Bijelic V, Borghese MM, Davis A, Reid S, Sangha G, Yeates KO, Tremblay MS, McGahern C, Belanger K, Barnes JD, Farion KJ, DeMatteo CA, Reed N, Zemek R; PERC PedCARE Concussion team. Is early activity resumption after paediatric concussion safe and does it reduce symptom burden at 2 weeks post injury? The Pediatric Concussion Assessment of Rest and Exertion (PedCARE) multicentre randomised clinical trial. Br J Sports Med. 2022 Mar;56(5):271-278. doi: 10.1136/bjsports-2021-105030. Epub 2021 Nov 26. PMID 34836880